CLINICAL TRIAL: NCT02976324
Title: The Effect of External Diaphragmatic Pacemaker on the Patients With Chronic Cor Pulmonale
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhang Xiangyu (Other)
Responsible Party: Sponsor-Investigator, Zhang Xiangyu, Director of Intensive care medicine, Tongji University
Organization: Tongji University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EDPCCP2016
Record Dates: First submitted 2016-11-08; First posted 2016-11-29 (Estimated); Last update posted 2017-10-23 (Actual); Status verified 2016-11

CONDITIONS: Chronic Cor Pulmonale
MeSH Terms: conditions — Pulmonary Heart Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- external diaphragmatic pacemaker group (Experimental): use the external diaphragmatic pacemakerI 9 counts per minute, with stimulate frequency 40 Hz
  Interventions: Device: external diaphragmatic pacemaker group
- control group (No Intervention): No inervention, just receive conventional therapy

INTERVENTIONS:
Device: external diaphragmatic pacemaker group — 9 counts per minute, with stimulate frequency 40 Hz
  Arms: external diaphragmatic pacemaker group

SUMMARY:
This study evaluates the effect of external diaphragmatic pacemaker on the patients with chronic cor pulmonale. Half of participants will receive external diaphragmatic pacemaker, while the other half will receive routine therapy.

DETAILED DESCRIPTION:
Investigate the effect of external diaphragmatic pacemaker on chronic cor pulmonale, the indicators include: respiratory muscle force, diaphragmatic degree of excursion and thickness, pulmonary artery pressure, respiratory distress, feeling of fatigue and quality of life, pulmonary function,NT-proBNP,PaO2 and PaCO2.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of chronic cor pulmonale and admit to hospital

Exclusion Criteria:

* pneumothorax or mediastinal emphysema
* active tuberculosis
* install a cardiac pacemaker
* acute cardiocerebrovascular events: acute myocardial infarction, acute myocarditis, severe arrhythmia, severe cerebrovascular accidents.
* pregnancies
* end-stage patients (expected survival time less than 6 months)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-11; Primary Completion 2017-05 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
cardiopulmonary function | 10 days
  six miunte walk test

SECONDARY OUTCOMES:
MIP | 10 DAYS
  MAX INSPIRATORY PRESSURE

CONTACTS AND LOCATIONS:
Overall Officials: xiangyu zhang, doctor, Principal Investigator — Tongji University
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided